CLINICAL TRIAL: NCT01028846
Title: Central Mechanisms That Regulate Glucose Metabolism in Humans
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: IRB approval expired 6/13/2023. Primary Completion Date and Study Completion Date updated after definitions were explained to PI/study team. Study never reached intended enrollment and will be categorized as terminated.
Sponsor: Meredith Hawkins (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); American Diabetes Association (Other)
Responsible Party: Sponsor-Investigator, Meredith Hawkins, Professor of Medicine, Albert Einstein College of Medicine
Organization: Albert Einstein College of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2006-414; R01DK069861 (NIH)
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Results first posted 2025-03-14 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes; Glucose Metabolism Disorders; Glucose, High Blood
Keywords: Type 2 Diabetes; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Diabetes Mellitus | interventions — Diazoxide

STUDY DESIGN:
Intervention Model Description: All participants received placebo or diazoxide in a randomized, double-blinded fashion.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diazoxide (Active Comparator): 4 mg/kg body weight total dosage administered orally during pancreatic clamp study
  Interventions: Drug: Diazoxide
- Placebo (Placebo Comparator): Saline administered orally during pancreatic clamp study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diazoxide — 4 mg/kg body weight total dosage administered orally
  Other Names: Proglycem
  Arms: Diazoxide
Drug: Placebo — Oral saline
  Arms: Placebo

SUMMARY:
Type 2 diabetes is a chronic condition that affects the ability of the body to regulate glucose (sugar). When glucose levels are low, the liver can make glucose to increase levels in the body. This important process is called endogenous glucose production (EGP). Previous studies suggest that the central nervous system (CNS), including the brain, helps to coordinate this process by communicating with the liver through potassium channels. Control of EGP can be impaired in people with type 2 diabetes, which may contribute to the high levels of glucose seen in these individuals.

The purpose of this study is to understand how activating these potassium channels in the control centers of the brain with a medication called diazoxide might inhibit the amount of glucose made by the liver. This is particularly important for people with diabetes who have very high production of glucose, which in turn causes hyperglycemia (high levels of sugar in the blood) that leads to diabetes complications.

DETAILED DESCRIPTION:
In this study, the investigators will study healthy participants through a procedure called a "pancreatic clamp" study. During the clamp procedure, glucose (a sugar) and insulin (a hormone produced in the pancreas that regulates the amount of glucose in the blood) are infused with an intravenous catheter, and blood samples are collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are found in the body and are related to glucose metabolism. Endogenous glucose production (the production of sugar by the liver) will be measured in patients given diazoxide (a medication that activates potassium channels in the brain that may affect glucose production in the liver through brain-liver signaling), compared with when a placebo is given.

All experiments will consist of 240 min insulin/somatostatin (250 μg/hr) infusions with replacement of glucoregulatory hormones (glucagon 1 ng/kg·min; growth hormone 3 ng/kg·min). Throughout the study, the plasma glucose concentration will be maintained at basal levels ( ~90 mg/dl). This will be attained by infusion of insulin at adequate rates to maintain normoglycemia without requiring glucose infusion. Primed continuous infusions of High-performance liquid chromatography-purified [3-3H]-glucose will be initiated at t=0 (21.6 μCi bolus, then 0.15 μCi/min), to measure glucose fluxes. All infusions will be stopped at t=240 min. From t=0 to t=240 min, blood samples will be obtained for determinations of plasma glucose, insulin, glucagon, C-peptide, cortisol, growth hormone, free fatty acids (FFA), glycerol, and lactate, and for 3-3H-glucose determinations.

This registration is exclusive to Aim 1 of the study protocol, which determined the effect of diazoxide on hepatic glucose production in nondiabetic, healthy, young individuals under fixed hormonal conditions. Euglycemic (90 mg/dl x 4 hours) pancreatic clamp studies (n= 10), with either saline or diazoxide infusion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Be no more than 140% of body weight
* No concurrent illnesses

Exclusion Criteria:

* No clinical history or laboratory evidence of hyperlipidemia (LDL cholesterol < 160 mg/dL)
* Clinical history of Hypertension
* Clinical history of Heart disease
* Clinical history of Cerebrovascular disease
* Clinical history of Seizures
* Clinical history of Bleeding disorders
* Clinical history of Muscle disease
* Smokers
* Mentally disabled persons
* Prisoners
* Pregnancy
* Clinical history of ethanol or drug or toxin exposure which could be associated with neuropathy
* Subjects incapable of giving voluntary informed consent
* History of bleeding disorder
* Clinical history of prolonged Prothrombin Time (PT) or Partial Thromboplastin Time

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2006-11-02 (Actual); Primary Completion 2007-12-05 (Actual); Study Completion 2007-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Hawkins, M.D., M.S., Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kishore P, Boucai L, Zhang K, Li W, Koppaka S, Kehlenbrink S, Schiwek A, Esterson YB, Mehta D, Bursheh S, Su Y, Gutierrez-Juarez R, Muzumdar R, Schwartz GJ, Hawkins M. Activation of K(ATP) channels suppresses glucose production in humans. J Clin Invest. 2011 Dec;121(12):4916-20. doi: 10.1172/JCI58035. Epub 2011 Nov 7. PMID 22056385

RESULTS

PARTICIPANT FLOW:
Groups:
- Diazoxide Followed by Placebo: Participants were initially administered 4 mg/kg body weight total dosage of diazoxide orally followed by saline orally after a two-week washout period.
  Diazoxide: 4 mg/kg body weight total dosage administered orally.
  Placebo: Oral saline
- Placebo Followed by Diazoxide: Participants were initially administered saline orally followed by 4 mg/kg body weight total dosage of diazoxide orally after a two-week washout period.
  Placebo: Oral saline
  Diazoxide: 4 mg/kg body weight total dosage administered orally
Period: 1st Intervention
Arm/Group | Diazoxide Followed by Placebo | Placebo Followed by Diazoxide
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Washout (~1 Month)
Arm/Group | Diazoxide Followed by Placebo | Placebo Followed by Diazoxide
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: 2nd Intervention
Arm/Group | Diazoxide Followed by Placebo | Placebo Followed by Diazoxide
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants were administered 4 mg/kg body weight total dosage of diazoxide orally followed by saline orally after a two-week washout period.
  Diazoxide: 4 mg/kg body weight total dosage administered orally.
  Placebo: Oral saline
Arm/Group | All Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.4 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Endogenous Glucose Production (EGP)
Description: Rate of EGP (a measure of the body's production of sugar) was measured using analysis of blood samples taken throughout the pancreatic clamp procedure under various treatment conditions (e.g., diazoxide or placebo) by monitoring changes in the level of a non-radioactive, naturally occurring form of glucose (sugar). Rates were summarized by treatment (Diazoxide or Placebo) in mg/kg/min sing basic descriptive statistics.
Time Frame: Final 60 minutes (t=180-240 minutes) of the pancreatic clamp, 6-7 hours after dosing
Measure: Mean (Standard Error); unit: mg/kg/min
Groups:
- Diazoxide: Participants were administered 4 mg/kg body weight total dosage of diazoxide.
  Diazoxide: 4 mg/kg body weight total dosage administered orally.
- Placebo: Participants were administered saline orally.
  Placebo: Oral saline
Arm/Group | Diazoxide | Placebo
Number analyzed (Participants) | 10 | 10
mg/kg/min | 1.15 (0.13) | 1.63 (0.17)

ADVERSE EVENTS:
Time Frame: Patients were assessed for up to 8 hours during two separate visits approximately 1 month apart.
Arm/Group | Diazoxide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diazoxide (N=10) | Placebo (N=10)
Mild Hypoglycemia (Asymptomatic) (Metabolism and nutrition disorders) | 1 | 0 — Grade 1. During the observation period following the pancreatic clamp, a glucose level was noted to be 56 mg/dL. Dextrose subsequently infused and rapidly brought glucose levels to within normal limits. Subject remained asymptomatic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes